CLINICAL TRIAL: NCT02873299
Title: High-Frequency Repetitive Transcranial Magnetic Stimulation of the Right Dorsolateral Prefrontal Cortex in Post Traumatic Stress Disorder
Brief Title: High-Frequency Repetitive Transcranial Magnetic Stimulation of the Right Dorsolateral Prefrontal Cortex in PTSD
Acronym: rTMS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2011.0025
Record Dates: First submitted 2014-09-30; First posted 2016-08-19 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: PTSD, Post Traumatic Stress Disorder
Keywords: PTSD, Post Traumatic Stress Disorder
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment as usual (No Intervention): Treatment as usual, wait list control group
- rTMS at 10Hz (Active Comparator): 10 Hz rTMS of the right dorsolateral prefrontal cortex
  Interventions: Other: 10 Hz rTMS of the right dorsolateral prefrontal cortex
- rTMS at 20Hz (Active Comparator): 20 Hz rTMS of the right dorsolateral prefrontal cortex
  Interventions: Other: 20 Hz rTMS of the right dorsolateral prefrontal cortex

INTERVENTIONS:
Other: 10 Hz rTMS of the right dorsolateral prefrontal cortex — Ten sessions of 10 Hz rTMS of the right dorsolateral prefrontal cortex
  Arms: rTMS at 10Hz
Other: 20 Hz rTMS of the right dorsolateral prefrontal cortex — Ten sessions of 20 Hz rTMS of the right dorsolateral prefrontal cortex
  Arms: rTMS at 20Hz

SUMMARY:
The purpose of this study is to compare two slightly different methods of transcranial magnetic stimulation (TMS) to treat Post Traumatic Stress Disorder (PTSD)

DETAILED DESCRIPTION:
This is a randomized single-blind pilot study investigating the efficacy of high-frequency repetitive transcranial magnetic stimulation (rTMS) applied to the right dorsolateral prefrontal cortex at either 10 Hz or 20 Hz as compared to a treatment as usual group for the treatment of Post Traumatic Stress Disorder (PTSD) symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Diagnosis of Post-Traumatic Stress Disorder as determined by the SCID
* CAPS score of at least 40
* Males or females between 18-65 years of age
* Willing to give up new psychotherapy or changes in psychiatric medications during the course of the TMS treatment.

Exclusion Criteria:

* Current primary Axis I disorder including Schizophrenia, Bipolar Disorder type I, Major Depressive Disorder
* Patients with HDRS score ≥ 18
* A metallic implant in cranium (except the mouth)
* Patients with severe or unstable medical conditions, which in the opinion of the investigator would interfere with their progress or safety
* ECT treatment within the last three months
* Patients with a history of epilepsy
* Patients with neurological disorder leading to increased intracranial pressure
* Participation in a new course of psychotherapy during the 24 days of the study
* A new psychiatric medication within 6 weeks of enrolling in the study
* Changes in psychiatric medication within 2 weeks of starting the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale , CAPS | day 10
  The CAPS is the gold-standard, semi-structured interview that corresponds to DSM-IV criteria for PTSD.

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist, PCL | week 24
  The PCL consists of 17 items measured on a 5-point Likert scale ranging from "not at all" to "extremely

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Capobianco, MD, DFAPA, Principal Investigator — NMCSD
Locations (1):
- NMCSD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No